CLINICAL TRIAL: NCT04840641
Title: Flucloxacillin as an Inducer of CYP-enzymes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: SignaTope GmbH, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AKF-396; 2020-004044-28 (EudraCT Number)
Record Dates: First submitted 2021-03-23; First posted 2021-04-12 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers; Drug Drug Interaction
Keywords: CYP enzymes; Induction of CYP enzymes
MeSH Terms: interventions — Floxacillin; Caffeine; efavirenz; Losartan; Omeprazole; Metoprolol; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): The investigators measure the baseline of flucloxacillin and cocktaildrugs.
- Flucloxacillin treatment (Experimental): The investigators measure the concentration of flucloxacillin after 9 and 27 days and the concentration of cocktaildrugs after 10 and 28 days.
  Interventions: Drug: Flucloxacillin

INTERVENTIONS:
Drug: Flucloxacillin — Healthy volunteers will take 2x500 mg flucloxacillin 3 times a day for 31 days. The investigators will measure the baseline concentration of the 6-cocktaildrugs and flucloxacillin before start of 31 days of flucloxacillin treatment. On day 9 and 27 the investigators will measure the concentration of flucloxacillin. On day 10 and 28 the investigators will measure the concentration of the 6 cocktaildrugs
  Other Names: Caffeine; Efavirenz; Losartan; Omeprazole; Metoprolol; Midazolam
  Arms: Flucloxacillin treatment

SUMMARY:
Worldwide there is an increase in antibiotic resistance which may have potential fatal long-term consequences. This is due to extensive use and sometimes misuse of antibiotics in the treatment of harmless infections.

The aim of this study is to investigate if treatment with flucloxacillin increases drug metabolism in healthy volunteers through induction of cytochrome P450 (CYP) enzymes, CYP1A4, CYP2B6, CYP2C9, CYP2C19, CYP2D6, and CYP3A4.

The hypothesis is based on an in vitro study showing that flucloxacillin activates a receptor (PXR) responsible for transcription of CYP enzymes.

Trial subjects will ingest flucloxacillin for 31 days and at day 10 and 28 ingest a cocktail of 6 drugs to determine if the CYP enzymes have been induced. Plasma and urine will be drawn over 72 hours to determine the concentration of the 6 drugs and their metabolites.

Change in flucloxacillin concentration will also be measured at day 9 and 27 to establish if flucloxacillin induces its own metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* The following data have to be in the normal range or only clinical insignificantly different from this: eGFR, ALAT, bilirubin, HbA1c, haemoglobin
* BMI 18.5 - 29.9 kg m-2
* Non-smoker (abstained from smoking minimum 2 weeks before the first study day and during the trial)
* Generally healthy
* Willing to give informed consent

Exclusion Criteria:

* Known sensitivity to any of the used drugs or any excipients listed in section 6.1 in the Summary of Product Characteristics (SmPC).
* Known allergy towards penicillin or cephalosporines
* Any of the following diseases (current or previous):

Heart disease, known family history of prolonged QTc interval, sudden death or conditions that might prolonged QTc-intervals, hypotension, severe disturbance of electrolyte balance e.g. hypokalemia or hypomagnesemia, myasthenia gravis, lung- or respiratory diseases, an anatomically abnormality of the respiratory tract, sleep apnea syndrome

- Intake of any significant prescription drugs, over-the- counter drugs, herbal drugs or dietary supplements. Contraindicated drugs include: Benzodiazepines, beta blockers, ergot alkaloids, herbal preparations containing St. John's wort, antiarrhythmics, neuroleptics, antidepressive agents, antibiotics, antifungal agents, non-sedating antihistamines, antimalarials, methadone, elbasvir, grazoprevir, nelfinavir cisapride, pimozide, bepridil

* Alcohol abuse or if the Danish Health Authority recommendation regarding alcohol intake has been exceeded 2 weeks before the first study day (men 14 units alcohol/week, women 7 units alcohol/week)
* Women who are breastfeeding
* Positive pregnancy test at inclusion screening or at any of the study days
* Participation in any other interventional trials

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Change in Area under curve (AUC) of midazolam | Baseline and day 28
  Change in the activity of the drug metabolizing enzyme CYP3A4

SECONDARY OUTCOMES:
Change in AUC of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in AUC of the metabolite of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in Peak Plasma concentration (Cmax) of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in Cmax of the metabolite of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in Time to reach Cmax (Tmax) of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in Tmax of the metabolite of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in Renal Clearence (CLr) of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in CLr of the metabolite of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in Elimination half-life (T1/2) of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in T1/2 of the metabolite of midazolam | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP3A4
Change in AUC of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in AUC of the metabolite of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in Cmax of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in Cmax of the metabolite of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in Tmax of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in Tmax of the metabolite of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in CLr of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in CLr of the metabolite of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in T1/2 of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in T1/2 of the metabolite of metoprolol | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2D6
Change in AUC of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in AUC of the metabolite of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in Cmax of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in Cmax of the metabolite of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in Tmax of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in Tmax of the metabolite of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in CLr of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in CLr of the metabolite of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in T1/2 of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in T1/2 of the metabolite of omeprazole | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C19
Change in AUC of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in AUC of the metabolite of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in Cmax of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in Cmax of the metabolite of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in Tmax of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in Tmax of the metabolite of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in CLr of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in CLr of the metabolite of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in T1/2 of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in T1/2 of the metabolite of losartan | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2C9
Change in AUC of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in AUC of the metabolite of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in Cmax of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in Cmax of the metabolite of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in Tmax of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in Tmax of the metabolite of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in CLr of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in CLr of the metabolite of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in T1/2 of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in T1/2 of the metabolite of efavirenz | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP2B6
Change in AUC of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in AUC of the metabolite of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in Cmax of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in Cmax of the metabolite of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in Tmax of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in Tmax of the metabolite of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in CLr of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in CLr of the metabolite of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in T1/2 of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in T1/2 of the metabolite of caffeine | Day 10 and 28
  Change in the activity of the drug metabolizing enzyme CYP1A2
Change in AUC of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in AUC of the metabolite of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in Cmax of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in Cmax of the metabolite of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in Tmax of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in Tmax of the metabolite of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in CLr of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in CLr of the metabolite of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in T1/2 of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin
Change in T1/2 of the metabolite of flucloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of flucloxacillin

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared due to general data protection regulation (GDPR).